CLINICAL TRIAL: NCT00570661
Title: Phase II, Open Label, International, Multicentre Clinical Trial to Investigate Safety and Efficacy of Oral ITF2357 in Patients With Active Systemic Onset Juvenile Idiopathic Arthritis (SOJIA)
Brief Title: Open Label, Multicentre Trial to Assess Safety and Efficacy of ITF2357 in Active Systemic Juvenile Idiopathic Arthritis
Acronym: SOJIA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Italfarmaco (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSC/05/2357/19
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Results first posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Active Systemic; Onset Juvenile Idiopathic Arthritis
MeSH Terms: interventions — givinostat hydrochloride; givinostat; Histone Deacetylase Inhibitors

STUDY DESIGN:
Masking Description: Not applicable. The study was open label.
Oversight: Data Monitoring Committee: No

ARMS (1):
- ITF2357 (Experimental): ITF2357 hard gelatine capsules were administered orally, in fed conditions, at the cumulative daily dose of 1.5 mg/kg achieved by administration of 0.75 mg/kg at 12-hour interval for 4 weeks initially. The doses of 1.5 mg/kg/day were achieved by administration of an appropriate number of capsules of definite strength (dose strengths of 7.5, 10, 12.5, 15, 20 mg and 50 mg).
  Treatment was further prolonged up to 12 weeks in total if so suggested by the observed benefits and the lack of treatment-limiting toxicity
  Interventions: Drug: ITF2357

INTERVENTIONS:
Drug: ITF2357 — ITF2357 orally administered at the cumulative daily dose of 1.5 mg/kg, achieved by administration of different dose strengths identifiable by different colours.
  Other Names: Givinostat, histone deacetylase inhibitor

SUMMARY:
This study has the following objectives:

Primary objective:

- To determine the safety and tolerability of oral ITF2357 in patients with active SOJIA with inadequate response or intolerance to standard therapy with oral steroids and methotrexate, with or without previously used biologic agents.

Secondary objectives:

* to evaluate the effect of ITF2357 on disease activity in patients with active SOJIA
* to investigate the possibility of steroid dose tapering in patients with active SOJIA during ITF2357 treatment
* to assess the effect of ITF2357 on levels of circulating cytokines
* to assess the pharmacokinetic properties of ITF2357

DETAILED DESCRIPTION:
The present study has been designed in order to evaluate safety and tolerability of ITF2357 in patients with active SOJIA with inadequate response or intolerance to standard therapy with oral steroids and methotrexate, with or without previously used biologic agents, and to have a preliminary evaluation of efficacy of ITF2357 in the treatment of SOJIA.

ITF2357 will be administered orally at the daily cumulative dose of 1.5 mg/kg: this dose in children/young adults is considered roughly equivalent to the dose of 1 mg/kg/day in adults, which so far has been proven to be free of any relevant safety concerns both in healthy volunteers and in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Established diagnosis of Systemic SOJIA according to ILAR criteria for at least six months before the study entry, with inadequate response or intolerance to standard therapy with oral steroids and/or methotrexate, with or without previously used biologic agents.
2. Active disease for at least one month prior to enrolment as defined by the following criteria:

   * Presence of arthritis plus at least one of the following:

     * Fever, defined as a body temperature >= 37,5 C degree at least once a day during at least five consecutive days or presence of typical SOJIA intermittent temperature chart
     * Rash, defined by presence of typical SOJIA salmon pink rash on the trunk and elsewhere during the febrile episodes
     * Serositis (pericarditis, pleuritis, peritonitis) confirmed by ultrasound and/or X-ray exploration or by presence of typical ECG findings in the case of pericarditis
     * Lymphadenopathy, defined by lymph nodes enlargement to 1,5 cm or more localized anywhere within the body, and/or hepatomegaly and/or splenomegaly, confirmed by ultrasound evaluation and established after comparison to age standards for organ size
     * ESR >= 20 mm/h (first hour) and/or CRP >= 10 mg/L. in the absence of arthritis, two definite or one definite and one probable diagnostic criteria plus ESR >=20 mm/h (first hour) and/or CRP >=10 mg/L
3. Age at enrolment between 2 and 25 years
4. Age at first SOJIA diagnosis < 16 years
5. Previously introduced standard treatment of disease with steroids without satisfactory effect and concomitant treatment with oral steroids at a dose equivalent to >= 0,2 mg/kg/day of prednisolone, unmodified for at least four weeks before patient's enrolment
6. In case of concomitant methotrexate treatment, it has to be on stable dose >= 10mg/m2 weekly for al least 4 weeks before pt enrollment
7. Previous treatment with biologics, if any, during at least three months without satisfactory effect or with drug intolerability, discontinued for at least the period specified below before patient's enrolment:

   * Two months for etanercept
   * Six months for infliximab
8. Other disease-modifying anti-rheumatic drugs possibly previously introduced have to be discontinued for a period of at least five half lives
9. Concomitant nonsteroidal anti-inflammatory drugs, if any, on a stable dose for at least four weeks before patient's enrolment
10. Female of childbearing potential, using safe contraceptive measures
11. Signed written informed consent before starting any study procedure

Exclusion Criteria:

1. Ongoing clinical relevant viral infection (eg.: Herpes Zoster, Ebstein barr, CMV, Systemic fungal infections or history of recurrent serious bacterial infection)
2. History of macrophage activation syndrome
3. Clinically significant illness i.e. any condition (including laboratory abnormalities) that in the opinion of the Investigator places the patient to unacceptable risk for adverse outcome if he/she were to participate in the study
4. Psychiatric illness/social situations that would limit compliance with study medication and protocol requirements
5. Congenital heart and/or central nervous system disorders
6. Inherited metabolic diseases
7. Positive serological testing for anti HCV, anti HIV and HBsAg (to be performed at screening)
8. Pregnant or lactating women
9. Presence of malignancy
10. Any previous evidence, irrespective of its severity, of coronary disease, cardiac rhythm abnormalities or congestive heart failure
11. QTc interval > 450 msec at screening evaluation
12. Serum magnesium and potassium below the LLN at screening
13. Unavoidable concomitant treatment with any drug known for potential risk of causing Torsades de Pointes

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2006-09-12 (Actual); Primary Completion 2008-08-25 (Actual); Study Completion 2013-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nemanja Damjanov, MD, PhD, Principal Investigator — Institute of Rheumatology Belgrade
Locations (5):
- Romania (2):
  - Clinica Institute Fundeni.Pediatric Clinic 258 Sos. Fundeni,, Bucharest
  - Clinical Emergency Children Hospital "M.S. Curie" Paediatric Clinic no. I 20 Ctin. Brancoveanu Bvd., 041451 Bucharest 4th district, Bucharest
- Serbia (3):
  - University Clinical Centre NisClinic of Paediatrics Department for Rheumatology Bul Dr Zoran Djindjica, Niš, Nis
  - Mother and Child Health Institute "Dr. Vukan Cupic" Clinic of Paediatrics Radoja Dakica, Belgrade, Novi Belgrade
  - Institute of Rheumatology Belgrade Resavska, Belgrade

REFERENCES:
- [Derived] Vojinovic J, Damjanov N, D'Urzo C, Furlan A, Susic G, Pasic S, Iagaru N, Stefan M, Dinarello CA. Safety and efficacy of an oral histone deacetylase inhibitor in systemic-onset juvenile idiopathic arthritis. Arthritis Rheum. 2011 May;63(5):1452-8. doi: 10.1002/art.30238. PMID 21538322
- [Derived] Vojinovic J, Damjanov N. HDAC inhibition in rheumatoid arthritis and juvenile idiopathic arthritis. Mol Med. 2011 May-Jun;17(5-6):397-403. doi: 10.2119/molmed.2011.00030. Epub 2011 Feb 4. PMID 21308151

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seventeen patients were screened and enrolled in the study
Pre-assignment Details: Patients with SOJIA according to the International League against Rheumatism criteria, established before the age of 16 y and for at least 6 mo before the study entry, having active disease for at least 1 mo while receiving more than 0.2 mg/kg/day prednisolone or equivalent steroid with/without concurrent methotrexate therapy (≥ 10 mg/m2 weekly).
Groups:
- ITF2357: ITF2357 hard gelatine capsules were administered orally, in fed conditions, at the cumulative daily dose of 1.5 mg/kg achieved by administration of 0.75 mg/kg at 12-hour interval for 4 weeks initially. The doses of 1.5 mg/kg/day were achieved by administration of an appropriate number of capsules of definite strength (dose strengths of 7.5, 10, 12.5, 15, 20 mg and 50 mg).
  Treatment was further prolonged up to 12 weeks in total if so suggested by the observed benefits and the lack of treatment-limiting toxicity
  ITF2357: ITF2357 orally administered at the cumulative daily dose of 1.5 mg/kg, achieved by administration of different dose strengths identifiable by different colours.
Period: Overall Study
Arm/Group | ITF2357
Started | 17
Completed | 10
Not Completed | 7
Not completed — Disease worsening | 5
Not completed — Unmet criterion of sufficient therapeutic response | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Safety population: all recruited patients who received at least one dose of the study medication.
Arm/Group | ITF2357
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.18 (5.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 11
Region of Enrollment [Number; unit: participants]
  Romania | 5
  Serbia | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Completing Week 12 of Treatment
Description: The primary endpoint describes the number of patients who has completed week 12 of treatment with ITF2357, both in the Per protocol (PP) population and in the Intention to treat (ITT) population.
  ITF2357 hard gelatine capsules were administered orally, in fed conditions, at the cumulative daily dose of 1.5 mg/kg achieved by administration of 0.75 mg/kg at 12-hour interval for 4 weeks initially. The doses of 1.5 mg/kg/day were achieved by administration of an appropriate number of capsules of definite strength. Treatment was further prolonged up to 12 weeks in total if so suggested by the observed benefits and the lack of treatment-limiting toxicity.
Time Frame: At week 12
Population: Per Protocol (PP) population: all patients who completed the study without any major deviations from the protocol procedures. Intent-To Treat (ITT) population: all recruited patients who received study medication and for whom at least one safety or efficacy measurement is available.
Measure: Count of Participants; unit: Participants
Groups:
- ITF2357 - PP Population: All patients in the study PP population (N=9) completed 12 weeks of treatment with ITF2357 according to the specifications of the protocol and thus reached the primary end-point of the study.
- ITF2357 - ITT Population: The analysis was repeated on the ITT population: 10 out of the 17 patients in the ITT population completed 12 weeks of treatment and reached the primary end-point of the study.
Arm/Group | ITF2357 - PP Population | ITF2357 - ITT Population
Number analyzed (Participants) | 9 | 17
Participants
  Completers | 9 | 10
  Non completers | 0 | 7

2. Secondary Outcome: JIA Outcome Core Set Variables - Patient Global Assessment
Description: Patient/parent global Visual Analogue Scale (VAS) is from 0 to 100. The lower the score, the better the outcome.
Time Frame: At pretreatment visit, at weeks 2, 4, 6, 8, 10 and 12 (End of treatment), 1 month and 3 months follow up (FU1, FU3) in the PP and ITT populations respectively.
Population: Per Protocol (PP) population: all patients who completed the study without any major deviations from the protocol procedures.
  Intent-To-Treat (ITT) population: all recruited patients who received study medication and for whom at least one safety or efficacy measurement is available. Nevertheless, data on Patient Global Assessment were available only on: n=16 at week 4 and FU1, n=14 at week 6, week 12 and FU3, and n=12 at week 8 and week 10. Other data are missing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ITF2357 - PP Population | ITF2357 - ITT Population
Number analyzed (Participants) | 9 | 17
units on a scale
  Pre-treatment | 48.00 (22.50) | 47.71 (21.45)
  Week 2 | 43.33 (21.15) | 42.47 (21.30)
  Week 4: number analyzed (Participants) | 9 | 16
  Week 4 | 21.22 (14.00) | 28.88 (22.48)
  Week 6: number analyzed (Participants) | 9 | 14
  Week 6 | 19.11 (15.00) | 22.36 (18.33)
  Week 8: number analyzed (Participants) | 9 | 12
  Week 8 | 17.22 (14.59) | 18.00 (13.99)
  Week 10: number analyzed (Participants) | 9 | 12
  Week 10 | 17.44 (13.28) | 22.33 (19.58)
  Week 12: number analyzed (Participants) | 9 | 14
  Week 12 | 19.11 (14.57) | 24.21 (20.89)
  FU1: number analyzed (Participants) | 9 | 16
  FU1 | 18.11 (15.53) | 26.56 (18.02)
  FU3: number analyzed (Participants) | 9 | 14
  FU3 | 15.38 (15.32) | 22.71 (17.85)

3. Secondary Outcome: JIA Outcome Core Set Variables - Physician Global Assessment
Description: Physician global Visual Analogue Scale (VAS) is from 0 to 100. The lower the score, the better the outcome.
Time Frame: as for outcome 2
Population: Per Protocol (PP) population: all patients who completed the study without any major deviations from the protocol procedures
  Intent-To Treat (ITT) population: all recruited patients who received study medication and for whom at least one safety or efficacy measurement is available. Nevertheless, data on Physician Global Assessment were available only on n=16 at week 4 and FU1, n=15 at FU3, n=14 at week 6 and week 12, n=12 at week 8 and week 10. Other data are missing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ITF2357 - PP Population | ITF2357 - ITT Population
Number analyzed (Participants) | 9 | 17
units on a scale
  Pretreatment | 48.00 (22.50) | 47.71 (21.45)
  Week 2 | 43.33 (21.15) | 42.47 (21.30)
  Week 4: number analyzed (Participants) | 9 | 16
  Week 4 | 21.22 (14.00) | 28.88 (22.48)
  Week 6: number analyzed (Participants) | 9 | 14
  Week 6 | 19.11 (15.00) | 22.36 (18.33)
  Week 8: number analyzed (Participants) | 9 | 12
  Week 8 | 17.22 (14.59) | 18.00 (13.99)
  Week 10: number analyzed (Participants) | 9 | 12
  Week 10 | 17.44 (13.28) | 22.33 (19.58)
  Week 12: number analyzed (Participants) | 9 | 14
  Week 12 | 19.11 (14.57) | 24.21 (20.89)
  FU1: number analyzed (Participants) | 9 | 16
  FU1 | 18.11 (15.53) | 26.56 (18.02)
  FU3: number analyzed (Participants) | 9 | 15
  FU3 | 15.38 (15.32) | 22.71 (17.85)

4. Secondary Outcome: JIA Outcome Core Set Variables - Number of Joints With Active Arthritis
Description: Number of active joints is from 0 to 75. The lower the score, the better the outcome.
Time Frame: as for outcome 2
Population: Per Protocol (PP) population: all patients who completed the study without any major deviations from the protocol procedures
  Intent-To Treat (ITT) population: all recruited patients who received study medication and for whom at least one safety or efficacy measurement is available. Nevertheless, data on N. joints with active arthritis were assessed only on: n=16 at week 4 and FU1, n=15 at FU3, n=14 at week 6 and week 12, n=12 at week 8 and week 10. Other data are missing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ITF2357 - PP Population | ITF2357 - ITT Population
Number analyzed (Participants) | 9 | 17
units on a scale
  Pretreatment | 9.33 (8.70) | 9.82 (9.11)
  Week 2 | 7.11 (8.62) | 8.41 (9.49)
  Week 4: number analyzed (Participants) | 9 | 16
  Week 4 | 3.78 (5.47) | 6.38 (9.26)
  Week 6: number analyzed (Participants) | 9 | 14
  Week 6 | 3.44 (5.29) | 3.57 (4.33)
  Week 8: number analyzed (Participants) | 9 | 12
  Week 8 | 3.67 (4.85) | 3.42 (4.29)
  Week 10: number analyzed (Participants) | 9 | 12
  Week 10 | 2.89 (4.54) | 2.75 (4.03)
  Week 12: number analyzed (Participants) | 9 | 14
  Week 12 | 3.44 (4.59) | 4.86 (4.74)
  FU1: number analyzed (Participants) | 9 | 16
  FU1 | 3.00 (4.50) | 3.88 (4.49)
  FU3: number analyzed (Participants) | 9 | 15
  FU3 | 3.33 (4.58) | 5.00 (6.05)

5. Secondary Outcome: JIA Outcome Core Set Variables - Number of Joints With Limitation
Description: Number of joints with limited range of motion is from 0 to 75. The lower the score, the better the outcome.
Time Frame: as for outcome 2
Population: Per Protocol (PP) population: all patients who completed the study without any major deviations from the protocol procedures
  Intent-To Treat (ITT) population: all recruited patients who received study medication and for whom at least one safety or efficacy measurement is available. Nevertheless, data on N. joints with limitations were available only on: n=16 at week 4 and FU1, n=15 at FU3, n=14 at week 6 and week 12, n=12 at week 8 and week 10. Other data are missing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ITF2357 - PP Population | ITF2357 - ITT Population
Number analyzed (Participants) | 9 | 17
units on a scale
  Pretreatment | 10.00 (9.53) | 11.59 (14.00)
  Week 2 | 8.56 (9.76) | 10.41 (14.42)
  Week 4: number analyzed (Participants) | 9 | 16
  Week 4 | 6.44 (7.20) | 7.44 (11.56)
  Week 6: number analyzed (Participants) | 9 | 14
  Week 6 | 5.78 (7.17) | 7.86 (11.91)
  Week 8: number analyzed (Participants) | 9 | 12
  Week 8 | 5.78 (6.63) | 4.67 (6.08)
  Week 10: number analyzed (Participants) | 9 | 12
  Week 10 | 5.22 (6.32) | 4.42 (5.65)
  Week 12: number analyzed (Participants) | 9 | 14
  Week 12 | 4.78 (5.65) | 8.79 (12.27)
  FU1: number analyzed (Participants) | 9 | 16
  FU1 | 5.00 (5.92) | 7.94 (12.22)
  FU3: number analyzed (Participants) | 9 | 15
  FU3 | 5.22 (5.70) | 7.20 (8.79)

6. Secondary Outcome: JIA Outcome Core Set Variables - CHAQ
Description: The Childhood Health Assessment Questionnaire (CHAQ) is from 0 to 3. For each of 8 section (Dressing and care, Getting up, Eating, Walking, Hygiene, Grasping, Catching, Activities) answers patient is getting 0,1,2 or 3 points (no difficulties, some difficulties, much difficulties, unable to do, respectively). The sum of points is then divided by 8 to get score 0 - 3. The lower the score, the better the outcome.
Time Frame: as for outcome 2
Population: Per Protocol (PP) population: all patients who completed the study without any major deviations from the protocol procedures
  Intent-To Treat (ITT) population: all recruited patients who received study medication and for whom at least one safety or efficacy measurement is available. Nevertheless, data on CHAQ were available only on: n=16 at week 4 and FU1, n=14 at weeks 6, 12 and FU3, n=12 at weeks 8 and 10. Other data are missing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ITF2357 - PP Population | ITF2357 - ITT Population
Number analyzed (Participants) | 9 | 17
units on a scale
  Pretreatment | 1.55 (0.54) | 1.75 (0.74)
  Week 2 | 1.13 (0.57) | 1.39 (0.87)
  Week 4: number analyzed (Participants) | 9 | 16
  Week 4 | 0.93 (0.55) | 1.23 (0.88)
  Week 6: number analyzed (Participants) | 9 | 14
  Week 6 | 0.75 (0.56) | 1.02 (0.82)
  Week 8: number analyzed (Participants) | 9 | 12
  Week 8 | 0.58 (0.50) | 0.85 (0.82)
  Week 10: number analyzed (Participants) | 9 | 12
  Week 10 | 0.55 (0.50) | 0.85 (0.87)
  Week 12: number analyzed (Participants) | 9 | 14
  Week 12 | 0.58 (0.41) | 0.95 (0.82)
  FU1: number analyzed (Participants) | 9 | 16
  FU1 | 0.56 (0.39) | 1.02 (0.93)
  FU3: number analyzed (Participants) | 8 | 14
  FU3 | 0.58 (0.51) | 0.85 (0.78)

7. Secondary Outcome: JIA Outcome Core Set Variables - ESR
Description: Measurements of erythrocyte sedimentation rate (ESR) were performed at the local laboratory cooperating with each study site.
Time Frame: as for outcome 2
Population: Per Protocol (PP) population: all patients who completed the study without any major deviations from the protocol procedures
  Intent-To Treat (ITT) population: all recruited patients who received study medication and for whom at least one safety or efficacy measurement is available. Nevertheless, data on ESR were available only on: n=16 at week 4 and FU1; n=13 at FU3, n=12 at week 8, n=10 at week 6 and n=8 at week 10. Other data are missing.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | ITF2357 - PP Population | ITF2357 - ITT Population
Number analyzed (Participants) | 9 | 17
mm/hr
  Pretreatment | 65.22 (23.05) | 62.71 (31.76)
  Week 2 | 53.44 (26.54) | 59.12 (30.90)
  Week 4: number analyzed (Participants) | 9 | 16
  Week 4 | 52.67 (22.66) | 59.50 (34.71)
  Week 6: number analyzed (Participants) | 6 | 10
  Week 6 | 57.67 (20.66) | 53.90 (22.35)
  Week 8: number analyzed (Participants) | 9 | 12
  Week 8 | 49.33 (33.78) | 49.92 (31.20)
  Week 10: number analyzed (Participants) | 6 | 8
  Week 10 | 58.33 (23.40) | 59.25 (23.35)
  Week 12 | 56.44 (40.76) | 54.14 (37.07)
  FU1: number analyzed (Participants) | 9 | 16
  FU1 | 39.89 (28.32) | 46.31 (28.30)
  FU3: number analyzed (Participants) | 7 | 13
  FU3 | 44.57 (25.00) | 41.00 (25.02)

8. Secondary Outcome: Overall SFS Results - Sum of First Five Variables and Sum of Last Five Variables
Description: Modified Systemic Feature Score (SFS) variables included:
  * temperature, rash, lymph nodes, liver and spleen size, and clinical evidence of serositis (clinical variables)
  * ESR, CRP, leukocyte count, haemoglobin, thrombocyte count (laboratory variables).
  Items in both sets of variables were scored as present (1) or not present (0) based on predefined criteria.
  SFS data were presented as the sum of the first 5 items and the sum of the last 5 items. Each sum could range from a minimum of 0 to a maximum of 5.
Time Frame: At pretreatment visit, at weeks 2, 4, 6, 8, 10 and 12 (End of treatment), 1 month follow-up (FU1) in the PP and ITT populations respectively.
Population: Per Protocol (PP) population: all pts who completed the study without any major protocol deviations
  Intent-To-Treat (ITT) population: all recruited pts who received medication for whom at least one safety or efficacy measurement is available. But, data on the sum of the first 5 variables were available on: n=16 at week 4; n=15 at FU1; n=14 at weeks 6, 12; n=12 at weeks 8, 10. Data on the sum of the last 5 variables were available on: n=14 at weeks 6, 12; n=12 at weeks 8, 10; n=16 at FU1.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ITF2357 - PP Population | ITF2357 - ITT Population
Number analyzed (Participants) | 9 | 17
score on a scale
  Sum of first 5 (clinical) variables - pre-treatment | 1.33 (0.71) | 0.94 (0.75)
  Sum of first 5 (clinical) variables - Week 2 | 0.44 (0.73) | 0.35 (0.61)
  Sum of first 5 (clinical) variables - Week 4: number analyzed (Participants) | 9 | 16
  Sum of first 5 (clinical) variables - Week 4 | 0.11 (0.33) | 0.31 (0.48)
  Sum of first 5 (clinical) variables - Week 6: number analyzed (Participants) | 9 | 14
  Sum of first 5 (clinical) variables - Week 6 | 0.11 (0.33) | 0.14 (0.36)
  Sum of first 5 (clinical) variables - Week 8: number analyzed (Participants) | 9 | 12
  Sum of first 5 (clinical) variables - Week 8 | 0.11 (0.33) | 0.17 (0.39)
  Sum of first 5 (clinical) variables - Week 10: number analyzed (Participants) | 9 | 12
  Sum of first 5 (clinical) variables - Week 10 | 0.11 (0.33) | 0.33 (0.65)
  Sum of first 5 (clinical) variables - Week 12: number analyzed (Participants) | 9 | 14
  Sum of first 5 (clinical) variables - Week 12 | 0.22 (0.44) | 0.29 (0.47)
  Sum of first 5 (clinical) variables - FU1: number analyzed (Participants) | 9 | 15
  Sum of first 5 (clinical) variables - FU1 | 0.22 (0.44) | 0.20 (0.41)
  Sum of last 5 (lab) variables - pretreatment | 4.33 (1.00) | 4.24 (1.15)
  Sum of last 5 (lab) variables - week 2 | 2.44 (1.42) | 2.65 (1.17)
  Sum of last 5 (lab) variables - week 4 | 2.11 (0.93) | 2.25 (1.18)
  Sum of last 5 (lab) variables - week 6: number analyzed (Participants) | 9 | 14
  Sum of last 5 (lab) variables - week 6 | 1.56 (1.33) | 1.93 (1.21)
  Sum of last 5 (lab) variables - week 8: number analyzed (Participants) | 9 | 12
  Sum of last 5 (lab) variables - week 8 | 2.00 (1.66) | 1.92 (1.44)
  Sum of last 5 (lab) variables - week 10: number analyzed (Participants) | 9 | 12
  Sum of last 5 (lab) variables - week 10 | 2.00 (1.58) | 2.08 (1.38)
  Sum of last 5 (lab) variables - week 12: number analyzed (Participants) | 9 | 14
  Sum of last 5 (lab) variables - week 12 | 1.89 (1.45) | 2.07 (1.27)
  Sum of last 5 (lab) variables - FU1: number analyzed (Participants) | 9 | 16
  Sum of last 5 (lab) variables - FU1 | 2.22 (1.92) | 2.56 (1.67)

9. Secondary Outcome: Number of Patients With Presence or Absence of Each Item for Modified Systemic Feature Score (SFS) - Temperature
Description: SFS variables included:
  1. temperature
  2. rash
  3. lymph nodes
  4. liver and spleen size
  5. clinical evidence of serositis (pericarditis, pleuritis or peritonitis)
  6. ESR
  7. CRP
  8. leukocyte count
  9. haemoglobin
  10. thrombocyte count
  Temperature was scored as present or not present according to the following criterion: body temperature ≥ 37.5 °C at least once a day during at least five consecutive days or presence of typical SOJIA intermittent temperature chart (patients' temperature chart analysis).
Time Frame: Pre-treatment, Weeks 4, 8, 12, and 1-month follow up
Population: Per Protocol (PP) population: all patients who completed the study without any major deviations from the protocol procedures.
  Intent-To Treat (ITT) population: all recruited patients who received study medication and for whom at least one safety or efficacy measurement is available. Nevertheless, data on T are available only on: n=16 at week 4; n=15 at FU1; n=14 at week 12; n=12 at week 8. Other data are missing.
Measure: Number; unit: participants
Arm/Group | ITF2357 - PP Population | ITF2357 - ITT Population
Number analyzed (Participants) | 9 | 17
participants
  Temp - Pretreatment - absence | 4 | 10
  Temp - Pretreatment - presence | 5 | 7
  Temp - Week 4 - absence: number analyzed (Participants) | 9 | 16
  Temp - Week 4 - absence | 8 | 12
  Temp - Week 4 - presence: number analyzed (Participants) | 9 | 16
  Temp - Week 4 - presence | 1 | 4
  Temp - Week 8 - absence: number analyzed (Participants) | 9 | 12
  Temp - Week 8 - absence | 8 | 10
  Temp - Week 8 - presence: number analyzed (Participants) | 9 | 12
  Temp - Week 8 - presence | 1 | 2
  Temp - Week 12 - absence: number analyzed (Participants) | 9 | 14
  Temp - Week 12 - absence | 7 | 11
  Temp - Week 12 - presence: number analyzed (Participants) | 9 | 14
  Temp - Week 12 - presence | 2 | 3
  Temp - FU1 - absence: number analyzed (Participants) | 9 | 15
  Temp - FU1 - absence | 7 | 12
  Temp - FU1 - presence: number analyzed (Participants) | 9 | 15
  Temp - FU1 - presence | 2 | 3

10. Secondary Outcome: Number of Patients With Presence or Absence of Each Item for Modified Systemic Feature Score (SFS) - Typical SOJIA Rash
Description: SFS variables included:
  1. temperature
  2. rash
  3. lymph nodes
  4. liver and spleen size
  5. clinical evidence of serositis (pericarditis, pleuritis or peritonitis)
  6. ESR
  7. CRP
  8. leukocyte count
  9. haemoglobin
  10. thrombocyte count
  Typical SOJIA is a salmon pink rash on the trunk during the febrile episodes.
Time Frame: Pre-treatment, Weeks 4, 8, 12, and 1-month follow up
Population: Per Protocol (PP) population: all patients who completed the study without any major deviations from the protocol procedures.
  Intent-To Treat (ITT) population: all recruited patients who received study medication and for whom at least one safety or efficacy measurement is available. Nevertheless, data on this outcome are available only on: n=16 at week 4 and FU1; n=14 at week 12; n=12 at week 8. Other data are missing.
Measure: Number; unit: participants
Arm/Group | ITF2357 - PP Population | ITF2357 - ITT Population
Number analyzed (Participants) | 9 | 17
participants
  Rash - Pretreatment - absence | 6 | 14
  Rash - Pretreatment - presence | 3 | 3
  Rash - Week 4 - absence: number analyzed (Participants) | 9 | 16
  Rash - Week 4 - absence | 9 | 16
  Rash - Week 4 - presence: number analyzed (Participants) | 9 | 16
  Rash - Week 4 - presence | 0 | 0
  Rash - Week 8 - absence: number analyzed (Participants) | 9 | 12
  Rash - Week 8 - absence | 9 | 12
  Rash - Week 8 - presence: number analyzed (Participants) | 9 | 12
  Rash - Week 8 - presence | 0 | 0
  Rash - Week 12 - absence: number analyzed (Participants) | 9 | 14
  Rash - Week 12 - absence | 9 | 14
  Rash - Week 12 - presence: number analyzed (Participants) | 9 | 14
  Rash - Week 12 - presence | 0 | 0
  Rash - FU1 - absence: number analyzed (Participants) | 9 | 16
  Rash - FU1 - absence | 9 | 16
  Rash - FU1 - presence: number analyzed (Participants) | 9 | 16
  Rash - FU1 - presence | 0 | 0

11. Secondary Outcome: Number of Patients With Presence or Absence of Each Item for Modified Systemic Feature Score (SFS) - Lymphadenopathy
Description: SFS variables included:
  1. temperature
  2. rash
  3. lymph nodes
  4. liver and spleen size
  5. clinical evidence of serositis (pericarditis, pleuritis or peritonitis)
  6. ESR
  7. CRP
  8. leukocyte count
  9. haemoglobin
  10. thrombocyte count
  Lymphadenopathy was scored as present or not present according to the following criterion: lymph node (nodes) enlargement to 1.5 cm or more, localized anywhere within the body.
Time Frame: Pre-treatment, Weeks 4, 8, 12, and 1-month follow up
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | ITF2357 - PP Population | ITF2357 - ITT Population
Number analyzed (Participants) | 9 | 17
participants
  Lymphadenopathy - Pretreatment - absence | 6 | 13
  Lymphadenopathy - Pretreatment - presence | 3 | 4
  Lymphadenopathy - Week 4 - absence: number analyzed (Participants) | 9 | 16
  Lymphadenopathy - Week 4 - absence | 9 | 16
  Lymphadenopathy - Week 4 - presence: number analyzed (Participants) | 9 | 16
  Lymphadenopathy - Week 4 - presence | 0 | 0
  Lymphadenopathy - Week 8 - absence: number analyzed (Participants) | 9 | 12
  Lymphadenopathy - Week 8 - absence | 9 | 12
  Lymphadenopathy - Week 8 - presence: number analyzed (Participants) | 9 | 12
  Lymphadenopathy - Week 8 - presence | 0 | 0
  Lymphadenopathy - Week 12 - absence: number analyzed (Participants) | 9 | 14
  Lymphadenopathy - Week 12 - absence | 9 | 14
  Lymphadenopathy - Week 12 - presence: number analyzed (Participants) | 9 | 14
  Lymphadenopathy - Week 12 - presence | 0 | 0
  Lymphadenopathy - FU1 - absence: number analyzed (Participants) | 9 | 16
  Lymphadenopathy - FU1 - absence | 9 | 16
  Lymphadenopathy - FU1 - presence: number analyzed (Participants) | 9 | 16
  Lymphadenopathy - FU1 - presence | 0 | 0

12. Secondary Outcome: Number of Patients With Presence or Absence of Each Item for Modified Systemic Feature Score (SFS) - Hepatomegaly and/or Splenomegaly
Description: SFS variables included:
  1. temperature
  2. rash
  3. lymph nodes
  4. liver and spleen size
  5. clinical evidence of serositis (pericarditis, pleuritis or peritonitis)
  6. ESR
  7. CRP
  8. leukocyte count
  9. haemoglobin
  10. thrombocyte count
  Hepatomegaly and/or splenomegaly was scored as present if confirmed by ultrasound evaluation and established after comparison to age standards for organ size.
Time Frame: Pre-treatment, Weeks 4, 8, 12, and 1-month follow up
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | ITF2357 - PP Population | ITF2357 - ITT Population
Number analyzed (Participants) | 9 | 17
participants
  Hepatomegaly - Pretreatment - absence | 8 | 16
  Hepatomegaly - Pretreatment - presence | 1 | 1
  Hepatomegaly - Week 4 - absence: number analyzed (Participants) | 9 | 16
  Hepatomegaly - Week 4 - absence | 9 | 16
  Hepatomegaly - Week 4 - presence: number analyzed (Participants) | 9 | 16
  Hepatomegaly - Week 4 - presence | 0 | 0
  Hepatomegaly - Week 8 - absence: number analyzed (Participants) | 9 | 12
  Hepatomegaly - Week 8 - absence | 9 | 12
  Hepatomegaly - Week 8 - presence: number analyzed (Participants) | 9 | 12
  Hepatomegaly - Week 8 - presence | 0 | 0
  Hepatomegaly - Week 12 - absence: number analyzed (Participants) | 9 | 14
  Hepatomegaly - Week 12 - absence | 9 | 14
  Hepatomegaly - Week 12 - presence: number analyzed (Participants) | 9 | 14
  Hepatomegaly - Week 12 - presence | 0 | 0
  Hepatomegaly - FU1 - absence: number analyzed (Participants) | 9 | 16
  Hepatomegaly - FU1 - absence | 9 | 16
  Hepatomegaly - FU1 - presence: number analyzed (Participants) | 9 | 16
  Hepatomegaly - FU1 - presence | 0 | 0

13. Secondary Outcome: Number of Patients With Presence or Absence of Each Item for Modified Systemic Feature Score (SFS) - Serositis
Description: SFS variables included:
  1. temperature
  2. rash
  3. lymph nodes
  4. liver and spleen size
  5. clinical evidence of serositis (pericarditis, pleuritis or peritonitis)
  6. ESR
  7. CRP
  8. leukocyte count
  9. haemoglobin
  10. thrombocyte count
  Serositis (pericarditis, pleuritis or peritonitis) was scored as present if confirmed by ultrasound and/or X-ray exploration or by the presence of typical ECG findings in the case of pericarditis.
Time Frame: Pre-treatment, Weeks 4, 8, 12, and 1-month follow up
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | ITF2357 - PP Population | ITF2357 - ITT Population
Number analyzed (Participants) | 9 | 17
participants
  Serositis - Pretreatment - absence | 9 | 16
  Serositis - Pretreatment - presence | 0 | 1
  Serositis - Week 4 - absence: number analyzed (Participants) | 9 | 16
  Serositis - Week 4 - absence | 9 | 15
  Serositis - Week 4 - presence: number analyzed (Participants) | 9 | 16
  Serositis - Week 4 - presence | 0 | 1
  Serositis - Week 8 - absence: number analyzed (Participants) | 9 | 12
  Serositis - Week 8 - absence | 9 | 12
  Serositis - Week 8 - presence: number analyzed (Participants) | 9 | 12
  Serositis - Week 8 - presence | 0 | 0
  Serositis - Week 12 - absence: number analyzed (Participants) | 9 | 14
  Serositis - Week 12 - absence | 9 | 13
  Serositis - Week 12 - presence: number analyzed (Participants) | 9 | 14
  Serositis - Week 12 - presence | 0 | 1
  Serositis - FU1 - absence: number analyzed (Participants) | 9 | 16
  Serositis - FU1 - absence | 9 | 16
  Serositis - FU1 - presence: number analyzed (Participants) | 9 | 16
  Serositis - FU1 - presence | 0 | 0

14. Secondary Outcome: Number of Patients With Presence or Absence of Each Item for Modified Systemic Feature Score (SFS) - Erythrocyte Sedimentation Rate (ESR)
Description: SFS variables included:
  1. temperature
  2. rash
  3. lymph nodes
  4. liver and spleen size
  5. clinical evidence of serositis (pericarditis, pleuritis or peritonitis)
  6. ESR
  7. CRP
  8. leukocyte count
  9. haemoglobin
  10. thrombocyte count
  At the pre-treatment visit ESR was scored as present or not present according to the following criterion: ESR considered as elevated if ≥ 20 mm/h (first hour)
  At the subsequent visits ESR was scored 0 (Not present) if decreased by at least 30% as compared to pre-treatment value or normalized (< 20 mm/h); score 1 (Present) if increased or decreased less than 30%.
Time Frame: Pre-treatment, Weeks 4, 8, 12, and 1-month follow up
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | ITF2357 - PP Population | ITF2357 - ITT Population
Number analyzed (Participants) | 9 | 17
participants
  ESR - Pretreatment - absence | 0 | 1
  ESR - Pretreatment - presence | 9 | 16
  ESR - Week 4 - absence: number analyzed (Participants) | 9 | 16
  ESR - Week 4 - absence | 2 | 5
  ESR - Week 4 - presence: number analyzed (Participants) | 9 | 16
  ESR - Week 4 - presence | 7 | 11
  ESR - Week 8 - absence: number analyzed (Participants) | 9 | 12
  ESR - Week 8 - absence | 4 | 4
  ESR - Week 8 - presence: number analyzed (Participants) | 9 | 12
  ESR - Week 8 - presence | 5 | 8
  ESR - Week 12 - absence: number analyzed (Participants) | 9 | 14
  ESR - Week 12 - absence | 3 | 5
  ESR - Week 12 - presence: number analyzed (Participants) | 9 | 14
  ESR - Week 12 - presence | 6 | 9
  ESR - FU1 - absence: number analyzed (Participants) | 9 | 16
  ESR - FU1 - absence | 4 | 6
  ESR - FU1 - presence: number analyzed (Participants) | 9 | 16
  ESR - FU1 - presence | 5 | 10

15. Secondary Outcome: Number of Patients With Presence or Absence of Each Item for Modified Systemic Feature Score (SFS) - C-reactive Protein (CRP)
Description: SFS variables included:
  1. temperature
  2. rash
  3. lymph nodes
  4. liver and spleen size
  5. clinical evidence of serositis (pericarditis, pleuritis or peritonitis)
  6. ESR
  7. CRP
  8. leukocyte count
  9. haemoglobin
  10. thrombocyte count
  At the pre-treatment visit CRP was scored as present or not present according to the following criterion: CRP considered as elevated if ≥ 10 mg/L.
  At the subsequent visits CRP was scored 0 (Not present) if decreased by at least 30% compared to pre-treatment value or normalized (< 10 mg/L); score 1 (Present) if increased or decreased less than 30%.
Time Frame: Pre-treatment, Weeks 4, 8, 12, and 1-month follow up
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | ITF2357 - PP Population | ITF2357 - ITT Population
Number analyzed (Participants) | 9 | 17
participants
  CRP - Pretreatment - absence | 0 | 0
  CRP - Pretreatment - presence | 9 | 17
  CRP - Week 4 - absence: number analyzed (Participants) | 9 | 16
  CRP - Week 4 - absence | 5 | 8
  CRP - Week 4 - presence: number analyzed (Participants) | 9 | 16
  CRP - Week 4 - presence | 4 | 8
  CRP - Week 8 - absence: number analyzed (Participants) | 9 | 12
  CRP - Week 8 - absence | 4 | 6
  CRP - Week 8 - presence: number analyzed (Participants) | 9 | 12
  CRP - Week 8 - presence | 5 | 6
  CRP - Week 12 - absence: number analyzed (Participants) | 9 | 14
  CRP - Week 12 - absence | 5 | 6
  CRP - Week 12 - presence: number analyzed (Participants) | 9 | 14
  CRP - Week 12 - presence | 4 | 8
  CRP - FU1 - absence: number analyzed (Participants) | 9 | 16
  CRP - FU1 - absence | 6 | 10
  CRP - FU1 - presence: number analyzed (Participants) | 9 | 16
  CRP - FU1 - presence | 3 | 6

16. Secondary Outcome: Number of Patients With Presence or Absence of Each Item for Modified Systemic Feature Score (SFS) - White Blood Cell (WBC)
Description: SFS variables included:
  1. temperature
  2. rash
  3. lymph nodes
  4. liver and spleen size
  5. clinical evidence of serositis (pericarditis, pleuritis or peritonitis)
  6. ESR
  7. CRP
  8. leukocyte count
  9. haemoglobin
  10. thrombocyte count
  At the pre-treatment visit WBC was scored as present or not present according to the following criterion: Leukocyte count considered as elevated if ≥ 12 x 103/μL.
  At the subsequent visits WBC was scored 0 (Not present) if decreased by 20% compared to pre-treatment value or normalized (< 12x103/μL); score 1 (Present) if increased or decreased less than 20%.
Time Frame: Pre-treatment, Weeks 4, 8, 12, and 1-month follow up
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | ITF2357 - PP Population | ITF2357 - ITT Population
Number analyzed (Participants) | 9 | 17
participants
  WBC - Pretreatment - absence | 2 | 4
  WBC - Pretreatment - presence | 7 | 13
  WBC - Week 4 - absence: number analyzed (Participants) | 9 | 16
  WBC - Week 4 - absence | 6 | 10
  WBC - Week 4 - presence: number analyzed (Participants) | 9 | 16
  WBC - Week 4 - presence | 3 | 6
  WBC - Week 8 - absence: number analyzed (Participants) | 9 | 12
  WBC - Week 8 - absence | 7 | 10
  WBC - Week 8 - presence: number analyzed (Participants) | 9 | 12
  WBC - Week 8 - presence | 2 | 2
  WBC - Week 12 - absence: number analyzed (Participants) | 9 | 14
  WBC - Week 12 - absence | 7 | 10
  WBC - Week 12 - presence: number analyzed (Participants) | 9 | 14
  WBC - Week 12 - presence | 2 | 4
  WBC - FU1 - absence: number analyzed (Participants) | 9 | 16
  WBC - FU1 - absence | 5 | 6
  WBC - FU1 - presence: number analyzed (Participants) | 9 | 16
  WBC - FU1 - presence | 4 | 10

17. Secondary Outcome: Number of Patients With Presence or Absence of Each Item for Modified Systemic Feature Score (SFS) - Haemoglobin (Hb)
Description: SFS variables included:
  1. temperature
  2. rash
  3. lymph nodes
  4. liver and spleen size
  5. clinical evidence of serositis (pericarditis, pleuritis or peritonitis)
  6. ESR
  7. CRP
  8. leukocyte count
  9. haemoglobin
  10. thrombocyte count
  At the pre-treatment visit Hb was scored as present or not present according to the following criterion: Haemoglobin considered as lowered if below 11g/dL.
  At the subsequent visits Hb was scored 0 (Not present) if increased by 20% compared to pre-treatment value or normalized (> 11 g/dL); score 1 (Present) if decreased or increased less than 20%.
Time Frame: Pre-treatment, Weeks 4, 8, 12, and 1-month follow up
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | ITF2357 - PP Population | ITF2357 - ITT Population
Number analyzed (Participants) | 9 | 17
participants
  Hb - Pretreatment - absence | 3 | 6
  Hb - Pretreatment - presence | 6 | 11
  Hb - Week 4 - absence: number analyzed (Participants) | 9 | 16
  Hb - Week 4 - absence | 4 | 6
  Hb - Week 4 - presence: number analyzed (Participants) | 9 | 16
  Hb - Week 4 - presence | 5 | 10
  Hb - Week 8 - absence: number analyzed (Participants) | 9 | 12
  Hb - Week 8 - absence | 4 | 6
  Hb - Week 8 - presence: number analyzed (Participants) | 9 | 12
  Hb - Week 8 - presence | 5 | 6
  Hb - Week 12 - absence: number analyzed (Participants) | 9 | 14
  Hb - Week 12 - absence | 4 | 6
  WBC - Week 12 - presence: number analyzed (Participants) | 9 | 14
  WBC - Week 12 - presence | 5 | 8
  Hb - FU1 - absence: number analyzed (Participants) | 9 | 16
  Hb - FU1 - absence | 4 | 8
  Hb - FU1 - presence: number analyzed (Participants) | 9 | 16
  Hb - FU1 - presence | 5 | 8

18. Secondary Outcome: Number of Patients With Presence or Absence of Each Item for Modified Systemic Feature Score (SFS) - Thrombocytes
Description: SFS variables included:
  1. temperature
  2. rash
  3. lymph nodes
  4. liver and spleen size
  5. clinical evidence of serositis (pericarditis, pleuritis or peritonitis)
  6. ESR
  7. CRP
  8. leukocyte count
  9. haemoglobin
  10. thrombocyte count
  At the pre-treatment visit thrombocyte count was scored as present or not present according to the following criterion: Thrombocyte count considered as increased if ≥ 400x103/μL.
  At the subsequent visits thrombocyte count was scored 0 (Not present) if decreased by 20% compared to pretreatment value or normalized (< 400x103/μL); score 1 (Present) if increased or decreased less than 20%.
Time Frame: Pre-treatment, Weeks 4, 8, 12, and 1-month follow up
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | ITF2357 - PP Population | ITF2357 - ITT Population
Number analyzed (Participants) | 9 | 17
participants
  Thrombocytes - Pretreatment - absence | 1 | 2
  Thrombocytes - Pretreatment - presence | 8 | 15
  Thrombocytes - Week 4 - absence: number analyzed (Participants) | 9 | 16
  Thrombocytes - Week 4 - absence | 9 | 15
  Thrombocytes - Week 4 - presence: number analyzed (Participants) | 9 | 16
  Thrombocytes - Week 4 - presence | 0 | 1
  Thrombocytes - Week 8 - absence: number analyzed (Participants) | 9 | 12
  Thrombocytes - Week 8 - absence | 8 | 11
  Thrombocytes - Week 8 - presence: number analyzed (Participants) | 9 | 12
  Thrombocytes - Week 8 - presence | 1 | 1
  Thrombocytes - Week 12 - absence: number analyzed (Participants) | 9 | 14
  Thrombocytes - Week 12 - absence | 9 | 14
  Thrombocytes - Week 12 - presence: number analyzed (Participants) | 9 | 14
  Thrombocytes - Week 12 - presence | 0 | 0
  Thrombocytes - FU1 - absence: number analyzed (Participants) | 9 | 16
  Thrombocytes - FU1 - absence | 6 | 9
  Thrombocytes - FU1 - presence: number analyzed (Participants) | 9 | 16
  Thrombocytes - FU1 - presence | 3 | 7

19. Secondary Outcome: Number of Patients With JIA Plus SFS Clinical Improvement
Description: Clinical improvement at week 2, 4, 6, 8, 10 and 12 was evaluated on the basis of JIA30, JIA50 and JIA70 plus SFS (two points decrease in SFS) as per protocol.
  Patients were considered as improved and with positive therapeutic response if 3 or more JIA Core Set Variables improved by 30% and no more than one worsened by 30%. JIA50 and JIA70 were defined as an improvement of 3 or more JIA Core Set Variables by 50% and 70%, respectively, and no more than 1 worsened by 30%. Additionally two points decrease in Systemic Feature Score were considered as disease improvement.
Time Frame: At weeks 2, 4, 6, 8, 10 and 12.
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | ITF2357 - PP Population | ITF2357 - ITT Population
Number analyzed (Participants) | 9 | 17
participants
  JIA30 plus SFS - W2 - Clinical improvement | 7 | 11
  JIA30 plus SFS - W2 - Absence of clinical improvement | 2 | 6
  JIA30 plus SFS - W4 - Clinical improvement | 8 | 12
  JIA30 plus SFS - W4 - Absence of clinical improvement | 1 | 5
  JIA30 plus SFS - W6 - Clinical improvement | 8 | 12
  JIA30 plus SFS - W6 - Absence of clinical improvement | 1 | 5
  JIA30 plus SFS - W8 - Clinical improvement | 8 | 11
  JIA30 plus SFS - W8 - Absence of clinical improvement | 1 | 6
  JIA30 plus SFS - W10 - Clinical improvement | 8 | 11
  JIA30 plus SFS - W10 - Absence of clinical improvement | 1 | 6
  JIA30 plus SFS - W12 - Clinical improvement | 8 | 10
  JIA30 plus SFS - W12 - Absence of clinical improvement | 1 | 7
  JIA50 plus SFS - W2 - Clinical improvement | 7 | 11
  JIA50 plus SFS - W2 - Absence of clinical improvement | 2 | 6
  JIA50 plus SFS - W4 - Clinical improvement | 8 | 10
  JIA50 plus SFS - W4 - Absence of clinical improvement | 1 | 7
  JIA50 plus SFS - W6 - Clinical improvement | 8 | 11
  JIA50 plus SFS - W6 - Absence of clinical improvement | 1 | 6
  JIA50 plus SFS - W8 - Clinical improvement | 8 | 10
  JIA50 plus SFS - W8 - Absence of clinical improvement | 1 | 7
  JIA50 plus SFS - W10 - Clinical improvement | 8 | 9
  JIA50 plus SFS - W10 - Absence of clinical improvement | 1 | 8
  JIA50 plus SFS - W12 - Clinical improvement | 8 | 9
  JIA50 plus SFS - W12 - Absence of clinical improvement | 1 | 8
  JIA70 plus SFS - W2 - Clinical improvement | 6 | 10
  JIA70 plus SFS - W2 - Absence of clinical improvement | 3 | 7
  JIA70 plus SFS - W4 - Clinical improvement | 8 | 10
  JIA70 plus SFS - W4 - Absence of clinical improvement | 1 | 7
  JIA70 plus SFS - W6 - Clinical improvement | 8 | 10
  JIA70 plus SFS - W6 - Absence of clinical improvement | 1 | 7
  JIA70 plus SFS - W8 - Clinical improvement | 8 | 9
  JIA70 plus SFS - W8 - Absence of clinical improvement | 1 | 8
  JIA70 plus SFS - W10 - Clinical improvement | 8 | 9
  JIA70 plus SFS - W10 - Absence of clinical improvement | 1 | 8
  JIA70 plus SFS - W12 - Clinical improvement | 8 | 9
  JIA70 plus SFS - W12 - Absence of clinical improvement | 1 | 8

20. Secondary Outcome: Number of Patients With Sufficient Therapeutic Response at Week 4 to Continue Treatment
Description: Therapeutic response at week 4 was considered sufficient by the Investigator if a decrease in Systemic Feature Score of 2 (at least one of the first five variables) and/or JIA30 response (or above: 50 or 70) was obtained.
Time Frame: At week 4
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | ITF2357 - PP Population | ITF2357 - ITT Population
Number analyzed (Participants) | 9 | 17
participants
  Therapeutic response | 8 | 11
  Absence of therapeutic response | 1 | 6

ADVERSE EVENTS:
Time Frame: At weeks 1, 2, 4, 6, 8, 10, 12 (end of treatment) and FU1 and FU3
Groups:
- IT2357 - Safety Population: Safety population: all recruited patients who received at least one dose of the study medication.
Arm/Group | IT2357 - Safety Population
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 2/17
Other Adverse Events (participants affected / at risk) | 14/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IT2357 - Safety Population (N=17)
Varicella (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IT2357 - Safety Population (N=17)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Fatigue (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (6)
Vomiting (Gastrointestinal disorders) | 1 (3)
Haematuria (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (3)
Influenza (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No